CLINICAL TRIAL: NCT05229380
Title: Pretympanoplasty Assessment of Patency and Mucociliary Function of Eustachian Tube
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Demiana Emad, demiana emad thabet, Assiut University
Other Study IDs: DEmadtympanoplasty
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- saccharin test: The patients with SPT less than 20 minutes are considered to have a normally functioning ET.
  The patients with SPT between 20- 45 minutes are considered to have a partial dysfunction of ET .
  The patients with SPT more than 45 minutes are considered to have a gross dysfunction of the ET .
  Interventions: Drug: Saccharin test
- methylene blue test: The patients with methylene blue clearance time less than 10 minutes are considered to have a normally functioning ET.
  The patients with methylene blue clearance time between10 to 20 minutes are considered to have a partial dysfunction of ET.
  The patients with methylene blue clearance time more than 20 minutes are considered to have a gross dysfunction of the ET .
  Interventions: Drug: Saccharin test

INTERVENTIONS:
Drug: Saccharin test — Saccharin is a nonnutritive sweetener. It has property of being inert to respiratory epithelium that is it does not hamper physiological mucus clearance of sino-nasal mucosa. Methylene blue is a chemical compound. It can be used to check patency of (ET). The dye, because of its liquid form, gravitates through the ET to the nasopharynx.
  Other Names: methyelne blue

SUMMARY:
The eustachian tube (ET) performs three primary functions: pressure equalisation between the nasopharyms and middle ear: clearance of mucus from the middle ear, and prevention of sound or fluid reflux from the nasopharynx(1) .In individuals suffering from custachian tube dysunction (ETD), the tube opening may be obstructed(2) resulting in the typical complaints of ear fullness, muffled hearing, or tinnitus(3). Less frequently, the ET may be permanently patulous, resulting in the symptoms of aural pressure or autophony (4). Adequate Eustachian tube function (ETF) is necessary for successful middle ear surgery. Studies of eustachian tube patency have been studied by the Politzer, Valsalva, and Toynbee maneuvers. In other cases it has been accomplished by testing air transport through the eustachian tube by tympanometry, sonotubometry, and air pressure equalization technique. However, these methods do not evaluate the drainage function (5). Saccharin is a nonnutritive sweetener. It has property of being inert to respiratory epithelium that is it does not hamper physiological mucus clearance of sino-nasal mucosa. It can be used to assess mucocilliary function of nasal mucosa, without itself hampering it. The saccharin test seems to provide adequate information of the mucociliary function and patency of the ET (6) . Methylene blue is a chemical compound. It can be used to check patency of (ET). The dye, because of its liquid form, gravitates through the ET to the nasopharynx. So the objective of the dye is to establish the anatomical presence or absence of tube patency.

DETAILED DESCRIPTION:
1. Full history taking, general and Complete otolaryngology examination to ride at any pathologies and focus of infection which could influence the result of tympanoplasty.
2. Audiological evaluation will be done for all patients both preoperatively and postoperatively
3. Computed Tomography scanning of the mastoids will be done for all cases to rule out mastoiditis of any type
4. Otoscopic examination size and site of perforation will be noted. The condition of middle ear mucosa, annulus, handle of malleus, and remnant of tympanic membrane (TM) will also be noted.
5. Diagnostic Nasal Endoscopy: detailed nasal examination will be carried out. The nasal findings and the condition of the ET orifice will be noted.
6. Saccharin test : Within two weeks before the surgery, the test will be performed. First, the taste response of patient to saccharin solution will br tested. With the patient seated and head tilted to the other ear , two drop of sterile sweety saccharin solution (one teaspoon saccharin granules dissolved in 10 ml sterile water) will placed in the middle ear through the TM defect by a dropper. The time required for the patient to taste the saccharin (ie, saccharin perception time [SPT]) will then measured.
7. Methylene Blue Test: Within two weeks before the surgery, the test will be performed. The nose is first prepared by applying a nasal pack soaked in a solution composed of mixture of xylometazoline hydrchloride 0.1% and xylocaine 10% (1:1) for 10 minutes. Then 0- degree sinscope (Karl storz, Germany) will passed through the nose till an adequate view of the nasopharyngeal opening of the ET is obtained. Two to three drops of sterile methylene blue dye will placed in the middle ear through the TM defect after tilting the patients head towards the opposite ear.
8. Within a week of evaluation of ETF, patients will be operated on for type 1 tympanoplasty after 3 weeks patients are reviewed for inspection of the operated ear. The second and third postoperative reviews will be done at 2 months and 6 months, respectively Patients were evaluated postoperatively by otoscopy, tympanometry, and audiometry.

ELIGIBILITY:
Inclusion Criteria:

1-Patients diagnosed with tubotympanic type of CSOM during quiescent stage (dry perforation).

Exclusion Criteria:

1. Active stage of tubotympanic CSOM (wet , discharging perforation).
2. Patients with atticoantral type of CSOM.
3. Patients with gross anatomical deformity or disease that can affect the result of tympanoplasty e.g cleft palate, severly deviated septum , adenoid, allergy , sinonasal polypi , otomycosis and presence of foci of infection.
4. Patients with previous ear surgery .
5. Patients with lost taste sensation .
6. Patients with sensorineural hearing loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data were collected and analyzed using SPSS (Statistical Package for the Social Science, version 20, IBM, and Armonk, New York). Continuous data were expressed in form of mean ± SD while nominal data were expressed in form of frequency (percentage). Frequency tables and charts were used .
  Chi²-test was used to compare the nominal data of different groups in the study. The level of confidence was kept at 95% hence a P value <0.05 indicated a significant association.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
out come of tympanoplasty | 2 years
  Tympanoplasty was considered successful if graft healing was noticed together with a mean of postoperative air bone gap of 20 dB or less at frequencies of 500,1000, 2000,4000 dB.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Prasad KC, Hegde MC, Prasad SC, Meyappan H. Assessment of eustachian tube function in tympanoplasty. Otolaryngol Head Neck Surg. 2009 Jun;140(6):889-93. doi: 10.1016/j.otohns.2009.02.015. Epub 2009 Apr 8. PMID: 19467410. — https://pubmed.ncbi.nlm.nih.gov/19467410/